CLINICAL TRIAL: NCT06931886
Title: Effects of Inspiratory Muscle Strength Training on Pulmonary Hypertension: A Six Week Study
Brief Title: Pulmonary Hypertension Inspiratory Training
Acronym: PHIT
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Elizabeth Fiona Bailey, PhD, Professor, University of Arizona
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00005343
Record Dates: First submitted 2024-12-09; First posted 2025-04-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-07

CONDITIONS: Pulmonary Hypertension
Keywords: Inspiratory Muscle Strength Training
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Intervention Model Description: Each individual enrolled will perform six weeks of inspiratory muscle strength training. There will be no control or sham group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Inspiratory Muscle Strength Training (Experimental): This group will perform inspiratory muscle strength training (~5 min/day) for 5 days a week for 6 weeks.
  Interventions: Other: Inspiratory Muscle Strength Training

INTERVENTIONS:
Other: Inspiratory Muscle Strength Training — Participants will be asked to inhale against a resistance. This resistance will be set to ~55% of their maximal inspiratory ability. Participants will complete 5 sets of 6 breaths (30 total) a day for 5 days a week for 6 weeks.
  Other Names: IMST; Resisted Breathing Training; Resisted Inspiratory Efforts

SUMMARY:
This study is examining the effects of six weeks of inspiratory muscle strength training (IMST) on outcomes related to pulmonary hypertension. This study leverages previous cardiopulmonary exercise test (CPET) results and a pre-existing upcoming CPET to examine the effects of IMST on cardiopulmonary pressures and exercise tolerance and ability.

DETAILED DESCRIPTION:
PH is a condition characterized by abnormally high blood pressure in the lungs (i.e., pulmonary arterial pressure), which impacts heart function and reduces exercise tolerance. This study will assess whether six weeks of a breathing exercise called IMST can improve heart and lung function as well as exercise capacity for individuals with PH.

For this study, patients will be asked to perform IMST for the six weeks prior to their next scheduled clinical standard of care assessment of their PH. The goal of this study is to determine whether IMST reduces pulmonary arterial pressure and improves exercise tolerance in individuals with PH. This study will be minimally invasive, as it simply adds a safe, well-tolerated, non-invasive respiratory training to the participants' standard of care and leverages their existing PH assessment data to evaluate the impact of IMST on PH.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with PH defined by clinical guideline criteria
* Must already be scheduled for a clinical assessment of their PH within 8 weeks of enrolling in the study.
* Must have undergone an assessment of their PH in the last 18 months with no major changes in PH management or medication within that period.

Exclusion Criteria:

* Current smoker or have smoked in the last 10 years
* Unable or unwilling to undergo routine functional testing of their PH (i.e., 6-minute walk distance).
* Presence of significant cardiovascular or respiratory conditions other than PH, including but not limited to:

  * Chronic obstructive pulmonary disease
  * Severe asthma
  * Severe ischemic heart disease
  * Left-sided heart failure
* History of a major cardiovascular event, such as a myocardial infarction or stroke, within the last 6 months
* Individuals with an implanted pacemaker or other significant cardiac devices
* History of neurological, respiratory, head and neck, or thoracic surgeries, or conditions such as a collapsed lung or perforated eardrum
* Pregnant individuals or those actively trying to become pregnant
* Individuals with any of the following: chronic laryngitis, chronic bronchitis, emphysema, pneumonia, tuberculosis, chronic cough, extremely high blood pressure (>170/100), neurological problems, scoliosis, organ transplants, HIV or other immunocompromising conditions, or autoimmune disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Estimated)
Dates: Start 2025-10-25 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Pulmonary arterial pressure | The data will be obtained from previous medical records of patient visits occurring up to 8 months prior to enrollment and at the end of treatment at 6 weeks post enrollment. .
  To be eligible for this study, patients must already have an upcoming invasive cardiopulmonary exercise test scheduled for assessment of their PH. Pulmonary arterial pressure will be obtained from this upcoming appointment as well as from previous medical records and an upcoming already scheduled assessment of pulmonary hypertension.
Cardiac Output | The data will be obtained from previous medical records of patient visits occurring up to 8 months prior to enrollment and at the end of treatment, which occurs 6 weeks post-initiation.
  This will be obtained as part of the usual standard assessment of pulmonary hypertension. Patients must already have this scheduled prior to enrollment in this study. Cardiac output, a measure of the volume of blood the heart pumps per minute, will be determined at rest and in response to exercise during the scheduled cardiopulmonary exercise test. This involves a graded maximal cycling protocol on a stationary bike, where resistance progressively increases until the patient reaches their maximum effort or exhaustion .
Maximal Oxygen Uptake | The data will be obtained from previous medical records of patient visits occurring up to 8 months prior to enrollment and at the end of treatment at 6 weeks post enrollment. .
  This will be obtained as part of the usual standard assessment of pulmonary hypertension. Patients must already have this scheduled prior to enrollment in this study. Maximal oxygen uptake, a measure of the body's maximum ability to take in, transport, and utilize oxygen during intense exercise, will be determined during the scheduled cardiopulmonary exercise test. This test involves a graded maximal cycling protocol on a stationary bike, where resistance progressively increases until the patient reaches their maximum effort or exhaustion. Throughout the test, patients will wear a mask that is used to analyze gas exchange.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Arizona, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided
These data will be preliminary and may be shared with other researchers with interest in PH.